CLINICAL TRIAL: NCT06941012
Title: Validation of α-synuclein Modifications in Parkinson's dIsoRder Evolution (VaMPiRE)
Brief Title: Validation of α-synuclein Modifications in Parkinson's dIsoRder Evolution
Acronym: VaMPiRE
Status: Recruiting | Type: Observational
Sponsor: Casa di Cura IGEA (Other)
Collaborators: Asociación Parkinson Madrid (Other); Aristotle University Of Thessaloniki (Other); Institute of Psychiatry and Neurology, Warsaw (Other); LINKCARE HEALTH SERVICES SL (Unknown); ALMAWAVE SPA (Unknown); European Brain Research Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 101156370
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease (PD)
Keywords: α-Synuclein
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson (PD)
  Interventions: Other: Blood draw for the laboratory assessment
- Non-PD controls
  Interventions: Other: Blood draw for the laboratory assessment

INTERVENTIONS:
Other: Blood draw for the laboratory assessment — Participants' clinical histories will be reviewed at T0 (baseline) and T1 (24 months). They will also undergo a clinical assessment at T0 and T1. The assessments will be tailored based on whether the participant belongs to the PD or non-PD group, as outlined below: • MDS-UPDRS + H&Y: Used to evaluate the neurological domain, applied to the PD group. • BERG: Used to assess balance and performance, applied to both PD and non-PD groups. • CIRS-G: Used to evaluate comorbidities, applied to both PD and non-PD groups. • PD-CRS: Used to assess cognitive function, applied to the PD group. • MMSE (temporal and spatial orientation only): Used to assess cognitive function, applied to both PD and non-PD groups. • PDQ-8: Used to evaluate quality of life, applied to the PD group. • PD-CFRS: Used for functional assessment, applied to the PD group. • GDS: Used to assess depression, applied to both PD and non-PD groups. Blood samples will be collected at T0 and T1, with 20 mL drawn per participant.
  Other Names: Neurologic evaluation

SUMMARY:
Parkinson's disease (PD) presents a complex challenge due to its progressive neurodegenerative nature, affecting various bodily systems. Despite decades of research, understanding its onset and progression remains unclear, complicating early diagnosis and treatment. Recent advances in PD pathophysiology suggest promising treatments to slow disease progression, yet reversing cellular degeneration remains elusive. With novel therapies emerging, the need for early detection tools is urgent. However, validated biomarkers for PD diagnosis are lacking, relying on subjective scales like Hoehn and Yahr or costly medical imaging techniques. The accumulation of misfolded α-Synuclein (α-Syn) proteins in PD pathology has sparked interest, but defining diagnostic roles requires further investigation. Recent findings of α-Syn in neuronal-derived extracellular vesicles (NDEVs) from PD patients suggest a potential for novel diagnostic methods. Our proposed project, VαMPiRE, aims to conduct a longitudinal study involving 600 PD and 600 non-PD participants using a cluster-adjusted case-control methodology, to explore α-Syn isoforms and related biomarkers in NDEVs for early PD detection.

We plan to develop and validate an innovative in-vitro diagnostic (IVD) test capable of detecting PD's earliest stages and estimating disease prognosis and progression. Utilizing AI models to generate data analysis algorithms and collaboration with leading analytical laboratories and IVD manufacturers, we aim to ensure the reliability and feasibility of the developed prototype. Through consortium efforts, we envision licensing the generated intellectual property to drive the commercialization of our results.

Two round of blood sample extractions will be performed within a 24-month gap to PD participants and a single baseline for non-PD controls. All participants will be regularly followed up during this 24-month period to monitor disease evolution and treatment, and non-PD controls developing the disease will be part of a third cohort (expected to be around 24 subjects according to 4% incidence) that will confirm the sensitivity of the test in asymptomatic subjects. The unique aspect of the project is that we anticipate being able to detect theses 4% of non-PD participants that will go on to develop the disease, therefore demonstrating the value of these biomarkers to identify PD early.

The prototype will be validated for its discriminative capacity, using the first baseline set of PD and non-PD samples, and for its ability to detect the PD-progression comparing baseline and 24-months data plus blood samples.

Improved early screening could allow for 270,000 new cases of PD to be detected earlier, improve the disease management of 9.4 M people currently diagnosed of PD and avoid losing a total of 5.8 million disability adjusted life years (DALYs) by 2028 leading also the development of better treatments.

DETAILED DESCRIPTION:
The VαMPiRE study (Validation of α-synuclein Modifications in Parkinson's dIsoRder Evolution) is a multicenter, longitudinal observational study in the context of European Grant Horizon Europe (101156370-2) and is designed to validate specific α-synuclein (α-Syn) isoforms and their post-translational modifications as biomarkers for the early detection and progression monitoring of Parkinson's disease (PD). The study addresses the critical unmet need for a cost-effective, non-invasive diagnostic method by combining innovative biochemical analyses, artificial intelligence (AI)-driven data models, and comprehensive clinical assessments. This effort aligns with emerging global priorities to enhance the early diagnosis and personalized treatment of neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* • For PD subjects

  * PD diagnosis according to MDS-UPDRS criteria and Hoehn and Yahr scale between I-IV (MED ON) for PD subjects
  * Willing to participate. Participation is always voluntary.
  * Willing and able to provide written informed consent to participate in the study or having a legal representative responsible for signing; the participant (or the legal representative) must understand the purpose, methods, and all information regarding the study.
  * For non-PD subjects
  * Normal neurological examination findings.
  * Medical record (recent and remote medical history) available and reviewable by clinicians during the entire study period.
  * Willing and able to provide written informed consent to participate in the study

Exclusion Criteria:

* • For PD and non-PD subjects

  * Clinically significant and severe cognitive decline and/or intellectual disability which can lead to impairment not caused by Parkinson's disease or any other disease that could better explain the patient's symptoms; The exclusion criteria involve neurological and neurodevelopmental disorders including disorders of the brain, spinal cord, peripheral nerve, and muscle (e.g. cerebral palsy, epilepsy [seizure disorders], stroke, intellectual disability, moderate to severe developmental delay, muscular dystrophy, or spinal cord injury).
  * Fever (Temperature 38.0 °C (tympanic)).
  * Acute infection (such as Flu, COVID-19) which could debilitate the patient and affect the data.
  * Individuals with concurrent infections requiring systemic antimicrobial and/or antiviral therapy at the pre-dose examinations (e.g. HepC, HIV, TB).
  * Life-threatening co-existing disease with life expectancy, which could lead to premature dropout.
  * Any other neurological or systemic conditions that could confound results.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will be conducted across five clinical sites, with each site contributing based on its recruitment capacity and resources.
  PD patients and non-PD controls will be recruited among similar characteristics. A matched case-control approach will be implemented to meet the study's objectives. Matching will be used to control for potential confounding factors. By pairing or grouping participants with PD (cases) and those without PD (non-PD controls) based on shared characteristics-such as age, gender, geographic location, and relevant comorbidities (e.g., type 2 diabetes, hypertension, anemia, gastrointestinal dysfunction, etc.)-we aim to reduce bias and enhance statistical efficiency in adjusted analysis. As it will be difficult to exactly match all cases with equivalent controls, we will use the stratification to cluster PD and non-PD participants so comparative analysis can be performed between PD and non-PD equivalent clusters. Each time a participant is recruited into PD, he/
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Quantification of α-Synuclein Isoforms (-140, -126, -112, -98) and Their SUMOylated Forms in NDEVs from Blood Samples | Baseline (T0) and 24 months post-enrollment (T1).
  The primary outcome measure involves the quantification of α-synuclein (α-Syn) isoforms (-140, -126, -112, -98) and their SUMOylated forms in neuronal-derived extracellular vesicles (NDEVs) isolated from blood samples. Advanced biochemical techniques, including lateral flow immunoassay coupled with digital readers, are employed for precise quantification. AI-driven data analysis evaluates correlations between biomarker levels and Parkinson's Disease (PD) progression.
  Clinical Implications:
  This outcome aims to validate α-Syn biomarkers for early PD diagnosis, offering a non-invasive, cost-effective alternative to current methods like DaT imaging. Reliable identification of α-Syn isoforms could improve early intervention strategies, slow disease progression, and support personalized treatment plans. Additionally, it could provide insights into disease mechanisms, enhancing future therapeutic developments and enabling scalable, accessible diagnostic solutions globally.

SECONDARY OUTCOMES:
Validation of AI-Generated predictive score for PD diagnosis | Baseline (T0), every 3 months through periodic surveys, and 24 months post-enrollment (T1).
  Development and validation of artificial intelligence (AI)-powered diagnostic algorithms utilizing multivariate biomarker data, clinical assessments, and demographic variables. The AI model generates a predictive score correlating α-Syn biomarker levels with disease onset, progression, and treatment response. The validation process evaluates the model's sensitivity, specificity, and predictive accuracy for Parkinson's Disease diagnosis.

OTHER OUTCOMES:
Longitudinal Assessment of Patient-Reported Quality of Life (QoL) Using PDQ-8 | Baseline (T0) and 24 months post-enrollment (T1).
  The Parkinson's Disease Questionnaire-8 (PDQ-8) is employed to assess changes in patient-reported quality of life (QoL) over the study period. It evaluates mobility, daily activities, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. Scores are analyzed to monitor disease burden and its correlation with α-Syn biomarker levels.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Feligioni, PHD, Study Chair — EBRI-European Brain Research Insitute; Elda Judica, MD, Principal Investigator — Casa di Cura IGEA
Locations (4):
- Aristotle University of Thessaloniki, Thessaloniki, Greece
- Casa di Cura Igea, Milan, Mi, Italy
- Instytut Psychiatrii I Neurologii, Warsaw, Poland
- Asociacion Parkinson Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes, demographic and baseline characteristics will be made available to qualified researchers upon reasonable request, following publication of study results. Data will be shared through appropriate data repositories and in compliance with applicable ethical and legal regulations. Via submission of a data access request to the study sponsor. Data will be shared through a secure institutional repository (e.g., Zenodo, ORE, EOSC).Key Exploitable Results will be disseminated through the Horizon Results Platform.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication of the main study results. For a period of 5 years following publication.

REFERENCES:
- See also: Related Info — https://www.vampire-eu.com/